CLINICAL TRIAL: NCT07232641
Title: Comparing Treatment Use, Retention, and Patient Outcomes Pre- and Post-implementation of Federal Policy Changes Regulating Buprenorphine and Methadone Treatment for Opioid Use Disorder
Brief Title: Impact of Federal and State Medications for Opioid Use Disorder (MOUD) Policy Changes During the Pandemic
Acronym: IMPACT
Status: Not yet recruiting | Type: Observational
Sponsor: Boston University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: H-46327; LTF-2024C2-39670 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute)
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Substance Use Disorders; Alcohol Use Disorder; Opioid Use Disorder
Keywords: Medications for opioid use disorder (MOUD)
MeSH Terms: conditions — Substance-Related Disorders; Alcoholism; Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- VA Patients with substance use disorder: Mutually exclusive groups of patients with OUD and AUD (and no co-occurring OUD), who will be matched 1:1 on age, gender, race, rural/urban residence, and state for the the pre (03/2016-02/2020) and post periods (03/2020-02/2024).

SUMMARY:
"Gold-standard" medications for opioid use disorder (MOUD) treatment combines FDA-approved medications, primarily methadone and buprenorphine, with behavioral therapies to provide "whole-patient" treatment. Prior to the pandemic, methadone and buprenorphine were subject to greater federal regulations than medications for other substance use disorders, including medication for alcohol use disorder (MAUD), which created barriers to MOUD initiation and retention. These barriers were exacerbated by physical distancing and diminished clinic capacities during the COVID-19 pandemic. To prevent healthcare disruption and expand access to MOUD treatment during the public health emergency, federal and state authorities implemented several MOUD policy changes during the pandemic to reduce barriers to MOUD initiation and retention, which subsequently became permanent.

This study is an evaluation of the impacts of these policies on treatment use, retention, and patient outcomes pre- and post-MOUD policy implementation.

DETAILED DESCRIPTION:
A mixed method study design will be implemented for this research study which has 3 specific aims.

Aim 1. Examine the long-term effects of MOUD policy changes on MOUD receipt, coverage, retention, and receipt of behavioral therapy, relative to commensurate measures among patients with AUD.

Aim 2. Examine the long-term effects of MOUD policy changes on outcomes for patients with OUD, including emergency department (ED) visits, inpatient hospitalization, substance use, relapse, and fatal and non-fatal overdoses, in contrast to pre-/post-period trends among our AUD comparison group.

Aim 3. Contextualize longitudinal results using qualitative methods to examine the impacts of MOUD policy changes from the perspectives of veteran patients with OUD, MOUD providers, and the Veteran's Health Administration Substance Use Disorder (VHA SUD) treatment leadership, and actors influencing the reach, effectiveness, adoption, implementation, and maintenance of MOUD policy changes.

For Aims 1 and 2, an observational cohort study will be conducted, using an interrupted time-series or difference-in-difference design to evaluate pre/post changes in treatment utilization and patient outcomes related to the nationwide MOUD policy changes introduced in 2020 expanding on access to MOUD treatment. The comparator for these analyses are patients with alcohol use disorder (AUD) for whom COVID-19 treatment disruptions applied but MOUD policies did not.

Data will be sourced from the Veteran's Health Administration Corporate Data Warehouse (CDW), including notes and Veteran's Administrations (VA) Mortality Data Repository and Community Care (CC) data. Aim 3 is a qualitative aim for which we will interview VA MOUD providers, VA substance use disorder treatment leadership, and VA patients with OUD.

ELIGIBILITY:
Inclusion Criteria:

* Substance use disorder (alcohol and/or opioid) documented in the Veteran's Health Administration Corporate Data Warehouse (CDW)

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A quasi-experimental and comparative interrupted time-series observational cohort study design will be used to compare trends across the pre- and post-MOUD policy change years, between mutually exclusive groups of patients with OUD and AUD (and no co-occurring OUD), who will be matched 1:1 on age, gender, race, rural/urban residence, and state for the pre (03/2016-02/2020) and post periods (03/2020-02/2024).
Sampling Method: Non-Probability Sample
Enrollment: 185810 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2029-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Change in MOUD/MAUD Receipt | 4 years pre/post policy change
  Based on Current Procedural Terminology (CPT) codes abstracted from the Veterans Administration VA Corporate Data Warehouse (CDW)
Change in MOUD/MAUD Coverage | 4 years pre/post policy change
  Based on Current Procedural Terminology (CPT) codes abstracted from the Veterans Administration VA Corporate Data Warehouse (CDW)
Change in MOUD/MAUD Retention | 4 years pre/post policy change
  Based on Current Procedural Terminology (CPT) codes abstracted from the Veterans Administration VA Corporate Data Warehouse (CDW)
Change in Behavioral Therapy Receipt | 4 years pre/post policy change
  Based on Current Procedural Terminology (CPT) codes abstracted from the Veterans Administration VA Corporate Data Warehouse (CDW)
Change in Behavioral Therapy Count | 4 years pre/post policy change
  Based on Current Procedural Terminology (CPT) codes abstracted from the Veterans Administration VA Corporate Data Warehouse (CDW)

SECONDARY OUTCOMES:
Change in any emergency department visits | 4 years pre/post policy change
  Receipt of any vs none emergency department visits based on Current Procedural Terminology (CPT) codes abstracted from the Veterans Administration VA Corporate Data Warehouse (CDW)
Change in the number of emergency department visits | 4 years pre/post policy change
  The count of emergency department visits based on Current Procedural Terminology (CPT) codes abstracted from the Veterans Administration VA Corporate Data Warehouse (CDW)
Change in any inpatient admissions | 4 years pre/post policy change
  Receipt of any vs none inpatient admissions based on Current Procedural Terminology (CPT) codes abstracted from the Veterans Administration VA Corporate Data Warehouse (CDW)
Change in the number of inpatient admissions | 4 years pre/post policy change
  The count of inpatient admissions based on Current Procedural Terminology (CPT) codes abstracted from the Veterans Administration VA Corporate Data Warehouse (CDW)
Change in any non-fatal Overdoses | 4 years pre/post policy change
  Defined as the presence of > International Classification of Diseases (ICD)-10 non-fatal overdose codes abstracted from the Veterans Administration VA Corporate Data Warehouse (CDW)
Change in the count of non-fatal Overdoses | 4 years pre/post policy change
  Based on non-fatal overdose codes abstracted from the Veterans Administration VA Corporate Data Warehouse (CDW)
Change in Fatal Overdoses | 4 years pre/post policy change
  Based on fatal overdose codes abstracted from the Veterans Administration VA Corporate Data Warehouse (CDW)
Change in Substance Use | 4 years pre/post policy change
  Documented in the electronic Health Record (EHR) and natural language processing large language models (NLP/LLM)
Change in Substance Use Relapse | 4 years pre/post policy change
  Documented in the electronic Health Record (EHR) and NLP/LLM

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Livingston, PhD, Principal Investigator — BUCA School of Medicine, Psychiatry and VA Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related parent grant. — https://clinicaltrials.gov/study/NCT03794986?term=NCT03794986&rank=1&tab=results